CLINICAL TRIAL: NCT04289428
Title: Evaluation of Novel Point of Care Hepatitis B Diagnostic Assays
Status: Withdrawn | Type: Observational
Why Stopped: Funding not awarded. A new study design and protocol have been submitted
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: VHCRP2001
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Diagnostics; HBV DNA; ALT; Point of care; Dried blood spot
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dried blood spot samples of capillary blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: Not currently on antiviral therapy for HBV and HBV DNA detectable
  Interventions: Diagnostic Test: Xpert® HBV DNA fingerstick point of care assay; Diagnostic Test: Point of Care ALT; Diagnostic Test: Xpert® HBV DNA point of care assay from dried blood spot
- B: Stable on HBV antiviral therapy for at least 3 months with HBV DNA < 20 IU/ml
  Interventions: Diagnostic Test: Xpert® HBV DNA fingerstick point of care assay; Diagnostic Test: Point of Care ALT; Diagnostic Test: Xpert® HBV DNA point of care assay from dried blood spot

INTERVENTIONS:
Diagnostic Test: Xpert® HBV DNA fingerstick point of care assay — Xpert® HBV DNA point of care assay from finger-stick whole blood
Diagnostic Test: Point of Care ALT — Point of Care ALT from finger-stick whole blood
Diagnostic Test: Xpert® HBV DNA point of care assay from dried blood spot — Xpert® HBV DNA point of care assay from dried blood spot

SUMMARY:
Evaluation of novel point of care Hepatitis B diagnostic assays.

DETAILED DESCRIPTION:
This study aims to evaluate the sensitivity of the following novel assays for evaluation of HBV infection and assessment of treatment eligibility;

* GeneXpert HBV DNA via Fingerstick testing,
* Dried Blood Spot based HBV DNA
* Point of care ALT.

ELIGIBILITY:
Inclusion Criteria:

1. Have voluntarily signed the informed consent form.
2. 18 years of age or older.
3. HBsAg positive
4. Part A: Not currently on antiviral therapy for HBV and HBV DNA detectable OR Part B: Stable on HBV antiviral therapy for at least 3 months with HBV DNA < 20 IU/ml

Exclusion Criteria:

1) Inability or unwillingness to provide informed consent or abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled into the study in two parts until the following sample sizes are met for the prospective samples Part A: At least 30 paired specimens of venous EDTA whole blood and DBS in treatment naive adults (HBV DNA detectable) Part B: At least 30 paired specimens of venous EDTA whole blood and DBS in HBV DNA undetectable adults on antiviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the Xpert® HBV DNA fingerstick point of care assay | Through study completion, an average of 1 year
  To evaluate the sensitivity and specificity of the Xpert® HBV DNA point of care assay from finger-stick whole blood samples compared to plasma samples collected via venipuncture and tested on the Roche COBAS AmpliPrep/COBAS TaqMan HBV (CAP/CTM HBV) V2 assay.

SECONDARY OUTCOMES:
Sensitivity and specificity of the point of care ALT | Through study completion, an average of 1 year
  To evaluate the sensitivity and specificity of the point of care ALT assay from finger-stick whole blood samples compared to standard of care ALT collected via venepuncture.
Sensitivity and specificity of the Xpert® HBV DNA point of care assay on dried blood spots | Through study completion, an average of 1 year
  To evaluate the sensitivity and specificity of the Xpert® HBV DNA point of care assay from dried blood spot samples compared to plasma samples collected via venipuncture and tested on the Roche COBAS AmpliPrep/COBAS TaqMan HBV (CAP/CTM HBV) V2 assay.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Matthews, MBBS, Principal Investigator — Kirby Institute
Locations (1):
- St. Vincent's Hospital Sydney, Darlinghurst, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No